CLINICAL TRIAL: NCT00155038
Title: Imaging Characteristics of Breast Cancer in Women Under 40 Years of Age
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700630
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2004-05

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Breast neoplasms; breast radiography; young women.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
To evaluate if there is any imaging characteristic of breast cancers in women younger than 40 years of age.

DETAILED DESCRIPTION:
In Western countries, breast cancer is the most commonly diagnosed cancer in women and breast cancer screening using mammography has reduced breast cancer mortality by 18-29%. In Taiwan, breast cancer is the second most common cancer in women and the Bureau of Health Promotion, Department of Health has started breast cancer screening using mammography in women between 50 and 69 years old since 2002, between 40 and 49 years old since early 2004. However, young women at 20 to 39 years of age have never been enrolled in the mass screening mammography program because of their relatively young age and mammographic findings of breast cancer in young women were seldom reported.Some authors found out that breast cancer in young women is more advanced and more often presents with a mass, has higher grade, more extensively proliferating and vessel invading disease when compared with those in older age groups. Most intraductal carcinomas (>80%) present as clustered microcalcifications on mammograms, and the sensitivity of mammography can be reduced in younger, denser breasts. Given these, mammography seems not to be a proper diagnostic tool for breast cancer women at a younger age. However, this presumption needs to be clarified since there are neither definite documented facts regarding breast cancer manifestation of young women on mammograms, nor documented sensitivity and false-negative rate of mammography in detecting of breast cancer among young women, at whom mammography is seldom used to be a diagnostic imaging tool. Our study is conducted to analyze the mammographic findings of breast cancers in young women between 20 and 39 years of age, regarding tumor size, location, major finding type, pathology type and grade. We will compare all of the above issues between younger age group and older age groups (40 to 49 and 50 to 69 years old).The breast ultrasound findings of the breast cancer among young women will be also compared with their corresponding mammographic findings, regarding the sensitivity, specificity, false-negative rate and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* 20-39 years women with breast cancers

Exclusion Criteria:

* pregnant women

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75
Dates: Start 1998-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Jane Wang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Colleoni M, Rotmensz N, Robertson C, Orlando L, Viale G, Renne G, Luini A, Veronesi P, Intra M, Orecchia R, Catalano G, Galimberti V, Nole F, Martinelli G, Goldhirsch A. Very young women (<35 years) with operable breast cancer: features of disease at presentation. Ann Oncol. 2002 Feb;13(2):273-9. doi: 10.1093/annonc/mdf039. PMID 11886005